CLINICAL TRIAL: NCT04656301
Title: Safety and Efficacy of Psilocybin for Body Dysmorphic Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: COMPASS Pathways (Industry); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Franklin Schneier, Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#7950
Record Dates: First submitted 2020-11-30; First posted 2020-12-07 (Actual); Results first posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-02

CONDITIONS: Body Dysmorphic Disorders
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Psilocybin (Experimental): A single dose of Psilocybin 25mg p.o.
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — A single dose of psilocybin 25 mg will be administered orally in the Biological Studies Unit of New York State Psychiatric Institute

SUMMARY:
In this pilot study 12 adult outpatients with body dysmorphic disorder that has not responded to at least one adequate trial of a serotonin reuptake inhibitor will be treated openly with a single oral dose of psilocybin. Followup visits to monitor safety and clinical outcome will be conducted over a 3 month period.

DETAILED DESCRIPTION:
In this pilot study, up to 12 adult outpatients with body dysmorphic disorder that has not responded to at least one adequate trial of a serotonin reuptake inhibitor will be treated openly with a single oral dose of psilocybin. Procedures will follow those previously established in depression studies of psilocybin. Patients will receive intensive preparation and support from two therapists, including 8-9 hours accompanying the patient on the day of medication administration in the Biological Studies Unit of New York State Psychiatric Institute. Followup visits to monitor safety and clinical outcome will be conducted at day 1, week1, and months 1,2, and 3 post-administration. Resting state function magnetic resonance imaging will be conducted prior to and one day after psilocybin administration to assess the effect of medication on brain circuits.

ELIGIBILITY:
Inclusion Criteria:

* Body dysmorphic disorder of at least moderate severity, non-delusional subtype, for >6 months
* History of intolerance of, or nonresponse to, a prior adequate trial of a serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI)
* Currently in psychotherapy (other than cognitive behavioral therapy (CBT) for body dysmorphic disorder

Exclusion Criteria:

* Current major depressive disorder of greater than moderate severity
* Other significant psychiatric or medical comorbidity or conditions that could interfere with safety of participation or interpretation of outcomes
* Use of: investigational medication within 3 months of baseline; depot antipsychotic within 6 months of baseline; serotonergic medication within 2 weeks of baseline (6 weeks for fluoxetine).
* Females who are pregnant, breastfeeding, or sexually active and not willing to use adequate contraception
* Enrollment in any investigational drug or device study in past 30 days
* Prior adverse effects from psilocybin

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Schneier, MD, Principal Investigator — Research Foundation for Mental Hygiene/NY State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, 1051 Riverside Drive, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu X, Zhang C, Hellerstein D, Feusner JD, Wheaton MG, Gomez GJ, Schneier F. Single-dose psilocybin alters resting state functional networks in patients with body dysmorphic disorder. Psychedelics (N Y). 2025;1(1):25-31. doi: 10.61373/pp024r.0028. Epub 2024 Sep 24. PMID 40458078

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Psilocybin
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Psilocybin
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.31 (8.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Body Dysmorphic Disorder Modification of the Yale-Brown Obsessive Compulsive Disorder Scale [Mean (Standard Deviation); unit: scale score] | 29.17 (4.60)

OUTCOME MEASURES:

1. Primary Outcome: Body Dysmorphic Disorder Modification of the Yale-Brown Obsessive Compulsive Disorder Scale
Description: The Yale-Brown Obsessive Compulsive Scale Modified for Body Dysmorphic Disorder (BDD-YBOCS) is a 12-item, semi-structured, rater-administered measure that assesses body dysmorphic disorder severity during the past week. Scores for each item range from 0 (no symptoms) to 4 (extreme symptoms); the total score ranges from 0 to 48, with higher scores reflecting more severe symptoms.
Time Frame: From baseline (day -1) up to 3 months post-dose
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psilocybin
Number analyzed (Participants) | 12
score on a scale | 18.42 (9.80)
Statistical Analysis 1: Comparison: Psilocybin; Test type: Superiority; p < 0.001, t-test, 2 sided; degrees of freedom = 1.92

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Psilocybin
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Psilocybin (N=12)
fatigue (General disorders) | 5 (5)
headache (Nervous system disorders) | 3 (3)
nausea (Gastrointestinal disorders) | 2 (2)
somnolence (Nervous system disorders) | 1 (1)
Lightheadedness (Nervous system disorders) | 1 (1)
spaciness (Nervous system disorders) | 1 (1)
insomnia (General disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
low libido (Reproductive system and breast disorders) | 1 (1)
emotional lability (Psychiatric disorders) | 1 (1)
visual hallucination (Psychiatric disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT04656301/Prot_SAP_000.pdf